CLINICAL TRIAL: NCT03437512
Title: Non-invasive Brain Stimulation in Adults Who Stutter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 paused human subjects research at study site, funding expired.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Emily O'Dell Garnett, Research Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00134495
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Stuttering, Developmental
Keywords: transcranial direct current stimulation; MRI; Speech; fluency; tDCS
MeSH Terms: conditions — Stuttering; Speech | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher who is not involved in any aspect of the study will randomize participants into the sham and active study arms using a minimization procedure. Allocation concealment will be achieved by assigning a unique 6-digit random code per participant, which will be provided to the researcher. The code is used to deliver stimulation. The participants and the researchers who deliver stimulation, assess outcomes, and analyze data will be masked to trial arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tDCS and fluency training (Experimental): Participants will receive anodal tDCS at 2milliampere (mA) intensity for 20 minutes during speech fluency training (5 consecutive days).
  Interventions: Device: Anodal tDCS; Behavioral: Fluency training
- Sham tDCS and fluency training (Sham Comparator): Participants will receive sham tDCS. Sham stimulation will involve 30 seconds of stimulation at the beginning of the 20 minutes of speech fluency training (5 consecutive days).
  Interventions: Behavioral: Fluency training; Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — 20 minutes of 2mA anodal stimulation.
  Arms: Active tDCS and fluency training
Behavioral: Fluency training — Speaking along with a metronome and/or speaking along with another person (choral speech) for 20 minutes
Device: Sham tDCS — For sham stimulation, current is ramped up and back down over 30 seconds.
  Arms: Sham tDCS and fluency training

SUMMARY:
Research studies in stuttering have shown that activity patterns in certain brain areas differ in people who stutter compared to people who do not stutter when speaking. The purpose of this study is to investigate how mild, non-invasive brain stimulation applied consecutively for five days affects speech relevant brain areas, which may in turn affect speech fluency and speaking-related brain activity in people who stutter.

ELIGIBILITY:
Inclusion Criteria:

* history of persistent developmental stuttering
* stuttering severity ranging from mild to very severe, specifically Stuttering Severity Instrument (SSI) total score of 20 (mild) or higher and stuttering rates of 3% or higher
* scores within 1 standard deviation of the norm on the standardized tests for the study

Exclusion Criteria:

* received any treatment for stuttering within the past year
* other neurological conditions such as Tourette's syndrome or post-traumatic stress disorder
* taking any medications/drugs that affect brain function
* history of past or current mental illness for example, schizophrenia that may affect brain development and function
* history of serious medical or neurological illness such as epilepsy and Parkinson's disease
* history of closed head injury (e.g., concussion)
* history of reading disorders
* hearing loss
* taking any medication, prescription or non-prescription with any psychotropic effects at the time of the study
* metal or electronic implants such as cochlear implants, and pacemakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily O Garnett, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were required to meet a certain stuttering severity status. Four participants who were enrolled did not meet the pre-assignment criteria and were thus not assigned to an arm.
Period: Randomized
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Started | 12 | 13
Completed | 12 | 11
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Received First tDCS Session
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Received Final tDCS Session
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Completed Study Follow up
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1
Not completed — Could not complete study due to COVID-19 research pause | 2 | 1

BASELINE CHARACTERISTICS:
Population: Includes all participants who were assigned to an arm and received the first intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.43 (8.14) | 23.31 (2.87) | 25.46 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Stuttering Severity [Mean (Standard Deviation); unit: percent] — Investigators will calculate the percentage of stuttered syllables (out of total syllables) in a speech sample. Decreased stuttered syllables represents better outcomes (greater reduction in stuttering).
  percent | 5.66 (3.23) | 9.72 (8.88) | 7.69 (6.06)
Overall Assessment of Speaker's Experience of Stuttering [Mean (Standard Deviation); unit: score on a scale] — The OASES is a standardized assessment of the functional impact of stuttering on a person's life. There are 4 sub-tests: general information about speech, your reactions to stuttering, communication in daily situations, quality of life. Each one has a score from 1 to 5 with regard to impact (1 least, 5 most negative impact). These are combined to give a total impact score between 1 and 5, with 5 representing the highest negative impact on person's life. The change on the total impact score will be used.
  score on a scale | 2.48 (0.58) | 2.67 (0.68) | 2.57 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Activation as Assessed by fMRI Images
Description: Investigators will use the fMRI images taken from before and after tDCS to determine if the treatment intervention contributed to any changes within brain regions associated with speech production. This will be measured by Blood-Oxygen-Level-Dependent (BOLD) signal change (arbitrary units). Images from scans are preprocessed. Changes in BOLD signal are modeled for contrasts within a group for [post-pre] and [follow up-pre] (e.g., active group reading condition post visit MINUS active group reading pre visit). Results are reported for reading condition.
Time Frame: Baseline, 1 week (post), 4 weeks (follow up)
Population: One subject assigned to the sham condition did not want to participate in the MRI but participated in every other aspect of the study. Additionally, 2 subjects assigned to active and 1 assigned to sham did not complete follow up MRI due to pandemic research pause. The MRI data from one subject in the active arm was corrupted and therefore not analyzable and was excluded from MRI results. Therefore [post-pre] includes 11 active and 10 sham, whereas [follow up-pre] includes 9 active and 9 sham.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Number analyzed (Participants) | 11 | 10
Percent signal change
  left supplementary motor area (SMA) (post-pre) | 1.39 (0.45) | 0.81 (0.47)
  left SMA (fol-pre): number analyzed (Participants) | 9 | 9
  left SMA (fol-pre) | 1.03 (0.49) | 0.9 (0.54)
  right SMA (post-pre) | -0.45 (0.48) | 0.49 (0.52)
  right SMA (fol-pre): number analyzed (Participants) | 9 | 9
  right SMA (fol-pre) | 0.86 (0.54) | 0.09 (0.35)
  left superior temporal gyrus (STG) (post-pre) | 1.43 (0.74) | 0.79 (0.75)
  left STG (fol-pre): number analyzed (Participants) | 9 | 9
  left STG (fol-pre) | 0.09 (0.53) | 0.57 (0.85)
  right STG (post-pre) | -0.63 (0.97) | 1.56 (1.39)
  right STG (fol-pre): number analyzed (Participants) | 9 | 9
  right STG (fol-pre) | 0.3 (1.07) | 0.83 (1.17)
  left putamen (post-pre) | 1.37 (0.66) | -0.31 (0.58)
  left putamen (fol-pre): number analyzed (Participants) | 9 | 9
  left putamen (fol-pre) | 2.42 (0.71) | -0.22 (0.59)
  right putamen (post-pre) | -1.01 (0.65) | -0.74 (0.67)
  right putamen (fol-pre): number analyzed (Participants) | 9 | 9
  right putamen (fol-pre) | 0.89 (0.69) | 0.06 (0.86)
  left inferior frontal gyrus (IFG) (post-pre) | 1.6 (0.94) | -0.33 (0.97)
  left IFG (fol-pre): number analyzed (Participants) | 9 | 9
  left IFG (fol-pre) | 0.23 (0.96) | 0.14 (0.74)
  right IFG (post-pre) | -0.48 (0.80) | 0.11 (0.65)
  right IFG (fol-pre): number analyzed (Participants) | 9 | 9
  right IFG (fol-pre) | -0.2 (0.80) | -0.2 (0.80)
  left premotor cortex (PMC) (post-pre) | 1.33 (0.91) | -0.15 (1.67)
  left PMC (fol-pre): number analyzed (Participants) | 9 | 9
  left PMC (fol-pre) | 0.68 (0.96) | 0.62 (1.11)
  right PMC (post-pre) | 0.31 (0.72) | 1.2 (0.93)
  right PMC (fol-pre): number analyzed (Participants) | 9 | 9
  right PMC (fol-pre) | 1.32 (1.01) | 1.01 (1.17)
Statistical Analysis 1: Comparison: Active tDCS and Fluency Training vs Sham tDCS and Fluency Training; Test type: Superiority; p < .001, t-test, 2 sided — familywise error rate (FWE) corrected to .05 with cluster threshold of 80 voxels

2. Primary Outcome: Change in Percentage of Stuttered Syllables Produced During Speech Sample
Description: Investigators will calculate the percentage of stuttered syllables (out of total syllables) in a speech sample. Decreased stuttered syllables represents better outcomes (greater reduction in stuttering).
Time Frame: Baseline, 1 week (post), 4 weeks (follow up)
Measure: Mean (Standard Deviation); unit: percent change in stuttered syllables
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Number analyzed (Participants) | 12 | 11
percent change in stuttered syllables
  % Change post | -1.82 (2.22) | 1.06 (2.02)
  % Change follow up | -1.03 (4.17) | 3.46 (5.47)
Statistical Analysis 1: Comparison: Active tDCS and Fluency Training vs Sham tDCS and Fluency Training; Analyses conduced with a mixed ANOVA, with between-subjects factor of group (active, sham) and two within-subjects factors: time (post, follow up) and speech task (reading, conversation); Test type: Superiority; p = .936, ANOVA — Interaction between visit and group

3. Secondary Outcome: Changes From Baseline on the Overall Assessment of Speakers Experience of Stuttering (OASES)
Description: The OASES is a standardized assessment of the functional impact of stuttering on a person's life. There are 4 sub-tests: general information about speech, your reactions to stuttering, communication in daily situations, quality of life. Each one has a score from 1 to 5 with regard to impact (1 least, 5 most negative impact). These are combined to give a total impact score between 1 and 5, with 5 representing the highest negative impact on person's life. The change on the total impact score will be used. Changes are shown in the table below by comparison between the measurements at the three points in time.
Time Frame: Baseline, 1 week (post), 4 weeks (follow up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
Number analyzed (Participants) | 12 | 11
score on a scale
  Pre | 2.48 (.61) | 2.67 (.75)
  Post | 2.34 (.55) | 2.56 (.78)
  Follow up | 2.35 (.57) | 2.59 (.88)
Statistical Analysis 1: Comparison: Active tDCS and Fluency Training vs Sham tDCS and Fluency Training; Test type: Superiority; p = .619, ANOVA — Interaction between visit and group

4. Other Pre Specified Outcome: Changes From Baseline on Rhythm Judgement Task
Description: Investigators will compare performance accuracy on a computerized rhythm judgement task from before and after tDCS to assess effects of tDCS. Improved accuracy reflects better performance.
Time Frame: Baseline, 1 week, 4 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes From Baseline on Tapping Tasks
Description: Investigators will compare performance on computerized tapping tasks from before and after tDCS to assess effects of tDCS.
Time Frame: Baseline, 1 week, 4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes From Baseline on Self-rated Measure of Speech Fluency
Description: Investigators will compare participant scores on a self-rated measure of speech fluency (1 = NO STUTTERING; 9 = EXTREMELY SEVERE STUTTERING) from before and after tDCS to assess effects of tDCS. Lower scores indicate improvement.
Time Frame: Baseline, 1 week, 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Active tDCS and Fluency Training | Sham tDCS and Fluency Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 12/12 | 10/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS and Fluency Training (N=12) | Sham tDCS and Fluency Training (N=11)
Headache (General disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 8 | 8
Tingling (Skin and subcutaneous tissue disorders) | 12 | 10
Warm sensation (Skin and subcutaneous tissue disorders) | 10 | 8
Sleepiness (General disorders) | 9 | 8
Trouble concentrating (General disorders) | 5 | 5
Acute mood change (General disorders) | 1 | 2
Fatigue (General disorders) | 6 | 4
Nervousness (General disorders) | 1 | 4
Changes in visual sensations (General disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Study was terminated early due to pandemic research pause, which resulted in fewer enrolled subjects than anticipated, which affected the number of subjects that could be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03437512/Prot_SAP_000.pdf